CLINICAL TRIAL: NCT01554475
Title: Use of Alternative Medicine Among Patients With Dementia and Mild Cognitive Dysfunction
Brief Title: Use of Alternative Medicine in Patients With Dementia and Mild Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: Kløveråsen Center for dementia, Bodø (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2011/1705(REK)
Record Dates: First submitted 2012-01-13; First posted 2012-03-15 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Dementia; Cognitive Impairment
Keywords: herbal drugs; dietary supplements; drug interactions
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
So far, no drugs have shown to stop or delay the pathological processes of dementia. Available pharmacological treatment includes a small number of drugs; cholinesterase inhibitors like donepezil, galantamine and rivastigmine, and the NMDA receptor antagonist memantine, all of which only affect the symptoms of the disease. At the same time, alternative medicines like herbal products and dietary supplements are often intensively marketed with the assertion of curative or alleviating effects on dementia. The documentation of clinical effects, side effects and the potential for interaction with prescribed drugs are, however, generally scarce. The aims of this study are to make a survey of the use of alternative medicine in patients with dementia and mild cognitive dysfunction attending the investigators out-patient dementia clinic, and to assess the interaction potential with the patient's other medications.

DETAILED DESCRIPTION:
Patients: All patients with a diagnosis of dementia under follow-up at the out-patient clinic are invited to participate, if giving a written consent.

Method: a semi-structured interview is undertaken by the doctor at the end of the consultation. Patients and their company are asked to name their alternative medicines (if any), for how long the products have been used, where and how they learned about the products, ant to tell about their experiences with the products (i.e if they have noticed effects or side-effects). After the consultation information of the the actual product's contents and properties are obtained and an assessment of possible interactions with the patient's other drugs (prescriptions and self-reported use of over-the-counter drugs) is made. Reported effects or side-effects are registered.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with dementia, under follow-up at Kløveråsen out-patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of patients taking alternative medicines | Up to 2 years
  The patient's use of alternative medicine(s) on a given point of time (the consultation date) as reported by the patient or by the next of kin who is the patient's companion during the consultation. The results will be presented as the number of patients taking alternative medicines

SECONDARY OUTCOMES:
Numbers of potential and clinical relevant interactions | Up to 2 years
  Assessment of the potential of interactions between the patient's alternative medicines and prescribed or over-the-counter drugs in use at the date of the consultation. The assessment will be based on data from litterature reports. Results will be presented as numbers of potential and clinical relevant interactions.
The patient's subjective experiences with alternative medicines | up to 2 years
  In the interview the patients will be asked to tell if they have experienced positive, negative, or no effects related to their use of alternative medicines. Results will be presented as number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Trude Giverhaug, PhD, Study Chair — University Hospital North-Norway
Locations (1):
- Kløveråsen, Bodø, Norway